CLINICAL TRIAL: NCT06572254
Title: Early Childhood Newborn Parenting Education Program at Primary Health Care Facilities of Pakistan: A Feasibility Study
Brief Title: ECD Newborn Parenting Education Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Global Affairs Canada (Other); Aga Khan Health Services (Other)
Responsible Party: Principal Investigator, Shelina Bhamani, Asst Professor, Lead Early Childhood Development and Program Director Outreach Education, Department of Obstetrics and Gynecology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8343
Record Dates: First submitted 2024-08-05; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Parenting
Keywords: Early childhood development; Responsive caregiving; Parenting

STUDY DESIGN:
Intervention Model Description: This study uses a parallel interventional design with two arms: an intervention group receiving a newborn parenting education program and a control group receiving no intervention. The primary aim is to compare parental confidence, feeding practices, teaching practices, and experiences between the two groups. Additionally, it assesses pre- and post-training experiences of nurses and healthcare providers and explores the readiness for large-scale implementation of the program in primary healthcare settings
Who Masked: Participant
Masking Description: Participants in the study will be randomly assigned to either the intervention arm, where they will receive the newborn parenting education program, or the control arm, where they will not receive any intervention. The participants will not be informed of their group allocation to minimize potential bias in their reporting of outcomes. Healthcare providers and researchers involved in the delivery of the intervention and data collection will be aware of the group allocations due to the practical requirements of implementing the education program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-study Pictorial Module (No Intervention): The control group will only be provided with a self-study pictorial module, and they will be tracked and requested to visit the center at the 6 months (child age) post-delivery. At 6 months, their data on responsive interactions, parenting confidence, and patient experience will be collected.
- Monthly Sessions and Self-study handouts (Experimental): The intervention will undergo a 6-month intervention consisting of 1 session at birth with a self-study manual, and 5 monthly sessions (once a month till the infant turns 6 months). At 6 months, they will also be assessed on the measures mentioned above.
  Interventions: Other: Early Childhood Development Newborn Parenting Education Program

INTERVENTIONS:
Other: Early Childhood Development Newborn Parenting Education Program — Investigators will be adapting the model used here at the tertiary care of newborn parenting which investogators have developed based on the nurturing care framework and keys to the caregiving framework. Both models have shown reliable evidence of their effectiveness.
  Other Names: Early Childhood Development Newborn Responsive Caregiving
  Arms: Monthly Sessions and Self-study handouts

SUMMARY:
Early childhood development: specifically the first 1000 days of life are of crucial importance. It sets the trajectory for the future and transgenerational health. Life of a neonate is influenced by several factors of which responsive caregiving is one of the most imperative facets. In the earliest days of life, the role of responsive caregiving is vital for the child's growing brain. Interactions between the primary caregiver and the neonate in early infancy period foster social and cognitive growth, build trust, provide sense of security, and helps build brain of the young child. In resource constraints areas, particularly in primary health care settings, there is a lack of initiatives to support responsive caregiving. The investigators intend to do an implementation adaptation and assessment of impact and efficacy of early childhood newborn parenting education program at primary health care facilities of Pakistan and Afghanistan. Investigators already have a structured program at our tertiary health care setting, with this project, investigators now intend to adapt it to primary care settings of Aga Khan Health Services Pakistan and Afghanistan a) explore the impact of newborn parenting education program on parental outcomes b) conduct training for health care providers and asses their pre-post knowledge and skills and c) explore systems readiness to scale up this program at national level. The expected outcome of this research is to build a proof of concept of this intervention in primary healthcare settings and disseminate its findings for a national level scale up and to advocate the importance of it to the government sector, civil society organization and funding agencies.

DETAILED DESCRIPTION:
The first 1000 days of life are critical to the growth and early brain development. Responsive caregiving lays the foundation of early childhood development and future acquisition of skills. Nurturing care provided by primary caregivers can activate different brain systems, allowing children to feel safe, form connections, and foster emotional and cognitive growth. A child's ability to adapt to adversity and stress in the future relies on a strong foundation of care provided in early childhood. The investigators also commit to be part of this movement and want to help realize the right of every child to survive and thrive, to build a more sustainable future for all. investigators are working on providing optimal care and wellbeing opportunities to the young children and this continuous and involved parenting support needs to start before birth and continue until the age of eight. The investigators will broadly take implementation research approach using different strategies for different aims. Hence for this research, investigators want to implement and adapt this same model in primary care settings of remote Pakistan and Afghanistan. The investigators have chosen Aga Khan Health Services Pakistan (AKHSP) and Aga Khan Health Services, Afghanistan (AKHSA), Foundation for Health and Empowerment (F4HE) field sites. The current research is also proposed in the same geographies that are part of F4HE, although F4HE has very strong implementation the research part is missing, so this research will fill the research gap and build knowledge on early childhood responsive caregiving in primary health care settings. AKHS has its primary care setup all over Pakistan and Afghanistan and the following BHCs will be chosen to implement this research and make the intervention sustainable.

ELIGIBILITY:
Inclusion Criteria:

1. Normal delivery
2. No underlying morbidities of the newborn
3. Are not living in ultra-poverty less than 15000/- total household income.

Exclusion Criteria:

1. Newborn or mother with underlying conditions or morbidities
2. Living under 15000 per month

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Scale | Baseline - At birth (1st Interaction)
  scale assesses an individual's perceived quality of life, including their physical health, psychological state, social relationships, and environmental factors. It evaluates how an individual's health status affects their overall well-being, happiness, and life satisfaction. The minimum value in the scale which is "1" indicates "very poor" while the maximum value which is "5" indicates "very good".
Karitine Parenting Confidence Scale | Through study completion, 6th month
  it consists of 15 items and is used by professionals. The items help explore caregivers' confidence in caring for their infants. It is a self-reported questionnaire and minimal clinical instructions are required to fill it. There are 4 Likert scale options out of which the minimum "0" indicates "No, hardly ever" while maximum is "3" which indicates "Yes, most of the time ". Parents scoring 39 or below indicate of experiencing low confidence while parents scoring 40 and above indicate high levels of confidence.
Responsive Interactions Scale | Through study completion, 6th month
  it consists of 15 items and is used by professionals. The items help explore caregivers' confidence in caring for their infants. It is a self-reported questionnaire and minimal clinical instructions are required to fill it. There are 4 Likert scale options out of which the minimum "0" indicates "No, hardly ever" while maximum is "3" which indicates "Yes, most of the time ". Parents scoring 39 or below indicate of experiencing low confidence while parents scoring 40 and above indicate high levels of confidence.
Caregiver Reported Early Development Instruments (CREDI) | Through study completion, 6th month
  The 20-item questionnaire is a brief version of the full Caregiver Reported Early Development Instruments, capturing essential developmental domains: cognitive, language, motor, and socio-emotional development. The minimum score is "0" while the maximum score is "20".

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Saleem, FCPS, Study Chair — Aga Khan University
Locations (2):
- Aga Khan Health Services, Kabul, Greater Kabul, Afghanistan
- Aga Khan Health Services, Chitral, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Investigators may not share the individual participant data but investigators plan to publish papers with partners from both countries and share the final results

REFERENCES:
- See also: A Packet for Parenting Education on Early Childhood Newborn Responsive Caregiving — https://www.aku.edu/mcpk/obs-gyn/Documents/ECD-English.pdf
- See also: "A Packet for Parenting Education on Early Childhood Newborn Responsive Caregiving — https://www.aku.edu/mcpk/obs-gyn/Documents/ECD-Urdu.pdf